CLINICAL TRIAL: NCT02143856
Title: A Randomized, Open-label, Two-way Cross-over Study to Determine the Oral Bioavailability of GLPG1205 After Single-dose Intake in Healthy Male Subjects as a Solid Formulation, With and Without Food
Brief Title: Oral Bioavailability of Solid Formulation of GLPG1205 With and Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GLPG1205-CL-102; 2013-004771-12 (EudraCT Number)
Record Dates: First submitted 2014-05-18; First posted 2014-05-21 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG1205

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 100 mg GLPG1205 fasted (Experimental): Single dose of 100 mg GLPG1205 as two capsules of 50 mg after an overnight fast
  Interventions: Drug: 100 mg GLPG1205
- 100 mg GLPG1205 fed (Experimental): Single dose of 100 mg GLPG1205 as two capsules of 50 mg exactly 30 minutes after the start of a high-fat, high-calorie breakfast
  Interventions: Drug: 100 mg GLPG1205

INTERVENTIONS:
Drug: 100 mg GLPG1205 — A single dose of 100 mg GLPG1205 administered as two capsules of 50 mg

SUMMARY:
The purpose of the study is to evaluate the amount of compound present in the blood (relative bioavailability) after a single oral administration of GLPG1205 given as a capsule formulation in fasted versus fed conditions in male healthy subjects.

Also, the safety and tolerability of a single oral dose of GLPG1205 given as a capsule formulation under fasted and fed conditions will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, age 18-50 years
* BMI between 18-30 kg/m2

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The amount of GLPG1205 in plasma | From predose up to 504 hours (Day 22) after study drug administration
  To characterize and compare the amount of GLPG1205 in plasma ( relative bioavailability) in male healthy subjects after a single administration of a capsule formulation in a fasted versus fed condition.

SECONDARY OUTCOMES:
The number of subjects with adverse events | From screening up to 28 (+/-2) days after last study drug administration
  To evaluate the safety and tolerability of a single dose of GLPG1205 administered as capsules fasted versus fed in male healthy subjects in terms of adverse events (AEs)
The number of subjects with abnormal laboratory parameters | From screening up to 28 (+/-2) days after last study drug administration
  To evaluate the safety and tolerability of a single dose of GLPG1205 administered as capsules fasted versus fed in male healthy subjects in terms of abnormal laboratory parameters
The number of subjects with abnormal vital signs | From screening up to 28 (+/-2) days after last study drug administration
  To evaluate the safety and tolerability of a single dose of GLPG1205 administered as capsules fasted versus fed in male healthy subjects in terms of abnormal vital signs
The number of subjects with abnormal electrocardiogram (ECG) | From screening up to 28 (+/-2) days after last study drug administration
  To evaluate the safety and tolerability of a single dose of GLPG1205 administered as capsules fasted versus fed in male healthy subjects in terms of abnormal electrocardiogram (ECG)
The number of subjects with abnormal physical examination | From screening up to 28 (+/-2) days after last study drug administration
  To evaluate the safety and tolerability of a single dose of GLPG1205 administered as capsules fasted versus fed in male healthy subjects in terms of abnormal physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Antwerp, Belgium